CLINICAL TRIAL: NCT01840553
Title: A Randomized Assessor-blinded Multicenter International Study Investigating Efficacy Patients Acceptance Safety and Tolerability of Sodium Phosphate Tablets Compared to Split Dose Polyethylene Glycol for Colon Cleansing Prior to Colonoscopy
Brief Title: Efficacy and Safety Study of Sodium Phosphate Tablets vs PEG for Bowel Cleansing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Mayoly Spindler (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICOL121; 2012-005115-13 (EudraCT Number)
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2013-11

CONDITIONS: Colon Cleansing
MeSH Terms: interventions — sodium phosphate; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- polyethylene glycol (Active Comparator): 4 Liters of PEG administered split in 2 doses
  Interventions: Drug: polyethylene glycol
- oral sodium phosphate tablets (Experimental): oral Sodium Phosphate tablets administered as 32 tablets (20+12) with 2 Liters of liquid
  Interventions: Drug: oral sodium phosphate tablets

INTERVENTIONS:
Drug: oral sodium phosphate tablets
  Arms: oral sodium phosphate tablets
Drug: polyethylene glycol
  Arms: polyethylene glycol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of sodium phosphate tablets compared to split dose of 4 liters of PEG used in adults for bowel cleansing prior to colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged from 18 to 75 years (included).
* Scheduled for a colonoscopy as an outpatient.
* Normal renal function

Exclusion Criteria:

* Having a disease or condition as follows:

  * repeated episodes of nausea and vomiting
  * abdominal pain due to severe infection or requiring surgery
  * clinically significant abnormal electrolytes values
  * congestive heart failure, unstable angina pectoris or recent myocardial infarction, percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass surgery within previous 3 months
  * known/suspected bowel obstruction, megacolon, ileus or intestinal perforation, or gastroparesis,
  * inflammatory bowel disease,
  * history of gastric stapling or bypass procedure or gastric retention
* Sodium phosphate preparation taken within the past three weeks prior to colonoscopy.
* Known allergy to any of the active ingredients or excipients of the study drugs.
* History of phenylketonuria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
overall quality of bowel cleansing | day 1

CONTACTS AND LOCATIONS:
Locations (19):
- France (8):
  - Hôpital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hopital Edouard Herriot, Lyon
  - Groupe Hospitalier Intercommunal Le Raincy-Montfermeil, Montfermeil
  - CHU Hotel Dieu, Nantes
  - Hopital l'Archet, Nice
  - CHU Cochin, Paris
  - Clinique Saint-Jean Languedoc, Toulouse
- Germany (4):
  - Sana Klinikum Lichtenberg, Berlin
  - Kreisklinik Biberach, Biberach
  - Klinikum Heidenheim, Heidenheim
  - Medizinische Klinik und Poliklinik II Munchen, München
- Spain (7):
  - Complejo Hospitalario de A Coruna, A Coruña
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de Fuenlabrada, Fuenlabrada
  - Hospital 12 de Octubre, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitarion Gregorio Maranon, Madrid
  - Clinica Universidad de Navarra, Pamplona

REFERENCES:
- [Derived] Chaussade S, Schmocker C, Toulemonde P, Munoz-Navas M, O'Mahony V, Henri F. Phosphate tablets or polyethylene glycol for preparation to colonoscopy? A multicentre non-inferiority randomized controlled trial. Surg Endosc. 2017 May;31(5):2166-2173. doi: 10.1007/s00464-016-5214-1. Epub 2016 Nov 18. PMID 27864718